CLINICAL TRIAL: NCT02437201
Title: Study of Liberty Program on Women's Health and Intimate Partner Violence: Multinational, Open, Randomised, Controlled Clinical Study
Brief Title: Study of Liberty Program on Women's Health and Intimate Partner Violence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Macmillan Research Group UK (Industry)
Collaborators: Goldington Family Center, UK (Unknown); Vinita Nursing Home, India (Other); Sonal Foundation, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Mac/NMP 1121
Record Dates: First submitted 2015-05-03; First posted 2015-05-07 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Violence Against Women

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liberty Group (Experimental): Weekly intensive support group for women with children who have suffered or are still suffering from domestic abuse (DA).
  Interventions: Behavioral: Liberty Program
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Liberty Program
  Arms: Liberty Group

SUMMARY:
Previous studies indicated high frequency of abuse in families and its consequences. Considering the importance of interventions such as educational interventions, in order to increase women's abilities to prevent abusive behaviors, the current research aims to determine the impact of an Liberty program on prevention of violence against women and propose solutions for less damages and consequences.

ELIGIBILITY:
Inclusion Criteria:

* Be married,
* Be under the aegis of Foundation at least for a year,
* Have at least one child.

Exclusion Criteria:

* Not participating in two educational sessions,
* Not being interested in continuing the cooperation.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Quality of Life measured by SF 36 Scale | Change from baseline in SF 36 Scale at 6 months

SECONDARY OUTCOMES:
Self-Esteem measured by Rosenberg Self-Esteem Questionnaire | Change from Baseline in Rosenberg Self-Esteem Questionnaire at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bharat B Chaudhari, MA, Study Director — Sonal Foundation, India; Paramjeet S Makkar, MD, Study Director — Vinita Nursing Home, India; Michael Howe, MA, Study Chair — Goldington Family Centre, UK; Avinash Mishra, MA, Study Director — Shanghai University, China
Locations (8):
- Liberty USA, Boston, Massachusetts, United States
- Liberty Australia, Melbourne, Australia
- Liberty China, Shanghai, Shanghai Municipality, China
- Liberty Europe, Athens, Greece
- India (2):
  - Sonal Foundation, Mahesāna, Gujarat
  - Vinita Nursing Home, Hindaun, Rajasthan
- Liberty Pakistan, Lahore, Punjaab, Pakistan
- Liberty Africa, Johannesburg, South Africa